CLINICAL TRIAL: NCT06076512
Title: Pain Clinic Provides Public Health and Safety Services
Brief Title: Pain Clinic Provides Public Health Safety
Status: Recruiting | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SalemAne2018 Pain HealthSafety
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Social Functioning; Addiction, Substance; Safety Issues; Road Injury; Patient Compliance; Chronic Pain
MeSH Terms: conditions — Social Adjustment; Substance-Related Disorders; Patient Compliance; Chronic Pain | interventions — Behavior Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult chronic pain patients: Adult chronic pain patients who received pain management and/or addiction therapy
  Interventions: Behavioral: Behavioral therapy

INTERVENTIONS:
Behavioral: Behavioral therapy — Behavioral and supportive therapy

SUMMARY:
Chronic pain is associated with psychological disorders; which may affect a patient's socioeconomic, legal, domestic, and employment situations. This prospective observational study evaluates the impact of pain management on patients' health, social, economic, and employment status. It explores the impact of pain clinic services on patients' mental health, family health, public health, road safety, addiction situation, public safety, injury rehabilitation and employment situation.

DETAILED DESCRIPTION:
Chronic pain is associated with many behavioral or psychological disorders. The psychological disorders may have negative impact on the patient's social, economic, health, legal, domestic, relationship and employment situations.

This prospective observational study evaluates the impact of pain management services on the patients' health, social, economic, and employment status. The clinical study explores the impact of pain clinic services on patients' mental health, childcare, family health, public health, road safety, addiction situation, public safety, injury rehabilitation, employment status and housing situation.

ELIGIBILITY:
Inclusion Criteria:

* adult chronic pain patients
* patients with psychosocial problems

Exclusion Criteria:

* pediatric patients
* patients with severe cognitive dysfunction

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult chronic pain patients who are undergoing treatment in a specialist pain clinic
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-02-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who had psychosocial problems | 12 months
  Percentage of patients who had psychosocial problems

CONTACTS AND LOCATIONS:
Overall Officials: Olu Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No